CLINICAL TRIAL: NCT06771466
Title: Patients' Satisfaction for Pain Control Modalities After Caesarean Section Using Erector Spinae Plain Block Vs Lateral Quadratus Lumborum Block. a Randomized Clinical Trial
Brief Title: Post-c-section Pain Control Satisfaction with Erector Spinae Simple Block Vs Lateral Quadratus Lumborum Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wael Sayed El Gharabawy (Other)
Responsible Party: Sponsor-Investigator, Wael Sayed El Gharabawy, assisstant professor of Anesthesia, Intensive care, and Pain management, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU R254/2024
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Satisfaction; Pain Management After Surgery
Keywords: nerve block, pain, opioids, patient satisfaction, cesarean section
MeSH Terms: conditions — Personal Satisfaction; Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: To investigate the difference in patient satisfaction following Erector spinae plane block (ESP) and Quadratus Lumborum block lateral approach after caesarean surgery, either alone or as part of multimodal analgesia.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient will be blind to the technique he will receive, and the care giver will be unaware of the block the patient being cared for received. Furthermore, the outcomes assessor, who is in charge of collecting the data, has no idea who received which block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bilateral Ultrasound-Guided Erector Spinae Plane Block (group E) (Active Comparator): those will receive Bilateral ultrasound-guided low thoracic Erector spinae plane block at a level of T9 with a total volume of 60 ml of bupivacaine 0.3% and Dexmedetomidine at a total dose of 0.5 mcg/kg
  Interventions: Procedure: Bilateral Ultrasound-Guided Erector Spinae Plane Block (group E)
- Bilateral Ultrasound-guided Quadratus Lumborum, Lateral approach (group Q) (Sham Comparator): Those patients will receive Bilateral ultrasound-guided Quadratus Lumborum, Lateral approach with a total volume of 60 ml of bupivacaine 0.3% and Dexmedetomidine at a total dose of 0.5 mcg/kg.
  Interventions: Procedure: Bilateral Ultrasound-guided Quadratus Lumborum, Lateral approach (group Q)

INTERVENTIONS:
Procedure: Bilateral Ultrasound-Guided Erector Spinae Plane Block (group E) — The curvilinear ultrasound transducer should be placed in a cephalocaudal orientation over the midline of the back at the desired level. The probe should then slowly be moved laterally until the transverse process is visible. The transverse process requires differentiation from the rib at that level. The transverse process will be more superficial and wider, while the rib will be deeper and thinner. Upon verification of the transverse process, the trapezius muscle, rhomboid major muscle (if performing at T5 level or higher), and erector spinae muscle should be identified superficial to the transverse process. The Tuohy needle should be inserted superior to the ultrasound probe using an in-plane approach in the cephalad to caudal direction.
  Arms: Bilateral Ultrasound-Guided Erector Spinae Plane Block (group E)
Procedure: Bilateral Ultrasound-guided Quadratus Lumborum, Lateral approach (group Q) — With the patient positioned in the lateral position, scanning is usually started at the mid-axillary line between the iliac crest and subcostal margin, moving the probe posteriorly until tapering of the three abdominal muscle layers and appearance of fascia transversalis and QL muscle are observed. The fascia transversalis usually appears as a hyperechoic layer, which forms a safe landmark to separate the muscle layers from the peri-nephric fat and the abdominal contents
  Arms: Bilateral Ultrasound-guided Quadratus Lumborum, Lateral approach (group Q)

SUMMARY:
The study will compare the difference between the patient's satisfaction after Erector spinae plane block (ESP) and Quadratus Lumborum block lateral approach after caesarean section alone or as part of multimodal analgesia.

The primary outcome is to test whether the type of plane block has an implication on the patients' satisfaction.

The secondary outcome is to test the difference between the two approaches on the hospital discharge

DETAILED DESCRIPTION:
The study will compare the difference between the patient's satisfaction after Erector spinae plane block (ESP) and Quadratus Lumborum block lateral approach after caesarean section alone or as part of multimodal analgesia. The primary outcome is to evaluate whether the type of plane block has an implication on the patients' satisfaction. The secondary outcome is to evaluate the difference between the two approaches on the hospital discharge.

Detailed Description IT is well Known that both Erector spinae plane block (ESP) and quadratus lumborum block are good modality for postoperative pain control after abdominal surgeries, this study will assess which one of both modalities is superior in achieving the patient's satisfaction after caesarean section. 1. INTRODUCTION: The goals for effective post-caesarean analgesia are interrelated and include allowing maternal bonding with her neonate, facilitating postoperative mobilization to reduce the risk of thromboembolism, preserving the ability for the mother to care for her infant, minimizing opioid use, and allowing safe breastfeeding with minimal transfer of analgesics to the neonate [1]. The options for post-caesarean delivery pain control include acetaminophen, non-steroidal anti-inflammatory drugs, intravenous opioids, fascial plane blocks, and neuro-axial opioids [1, 2]. Efforts to reduce the doses of opioids prescribed after CD, both in the hospital and after discharge, are increasing. The lowest effective dose of any opioid should be used to minimize breast milk transfer and associated neonatal sedation. Neuraxial opioids are preferred to other routes of administration, when possible, to minimize maternal blood and breast milk levels [3]. If opioids are required, breastfeeding should ideally start just prior to opioid administration, as the drug concentration in breast milk rises and falls in parallel with maternal plasma levels [3]. Highly protein-bound medications such as nonsteroidal anti-inflammatory drugs (NSAIDs) and local anesthetics transfer less readily into breast milk than opioids and other lipophilic drugs [4]. A reported advantage of QL blocks is the possibility of providing better visceral analgesia compared with TAP blocks. However, the literature on the relative benefits of QL versus TAP blocks and other blocks for post-CD analgesia is conflicting. However, QL blocks can result in lower extremity weakness, particularly for the variants that involve more central injection of LA as in anterior QL [5]. Available literature regarding the use of other nerve blocks (e.g., ESP, ilio-inguinal ilio-hypogastric [IIH], transversalis fascia plane, QL blocks) has been described but is limited regarding the analgesic effect, duration of action, quality of recovery and the relation to each other. [6,7]. It is well known that dermatomal coverage from ESP blocks depends on the volume and dose of local anesthetic administered. Blocks placed at low thoracic levels (e.g., T9 to 10) should provide appropriate coverage for low transverse incision for CD.

2. AIM/OBJECTIVES To study the difference between the patient's satisfaction after Erector spinae plane block (ESP) and Quadratus Lumborum block lateral approach after caesarean section alone or as part of multimodal analgesia. The primary outcome is to assess whether the type of the plane block has an implication on the patients' satisfaction. The secondry outcome is to assess the difference between the two approaches on the hospital discharge.

3. METHODOLOGY: Patients and Methods, Subjects and Methods, Material and Methods • Type of Study: Randomized clinical trial Study Setting: Obstetric and gynecological hospital, Faculty of medicine, Ain Shams university. • Study Period: 6 months • Study Population: Inclusion Criteria: • Parturient female • Scheduled for elective caesarean section Exclusion Criteria: • Known allergy to any of the medication used • Patients refused to participate in the study • Patients with emergency section • Patients with Bleeding disease • Patients with postpartum hemorrhage

• Sampling Method: The patients will be randomly divided into two equal groups; randomization will be done by computer-generated number lists. ALL the patients will receive spinal anesthesia after proper sterilization of the back with betadine, 2.5 ml of heavy Bupivacaine 0.5%, together with twenty-five micrograms of fentanyl at the level of L 4-5. The block was maintained at level T4. The patients will be divided into two groups: Group E includes sixty-three women; those will receive an ultrasound-guided low thoracic Erector spinae plane block at level of T9 with a total volume of 60 ml of bupivacaine 0.3% and Dexmedetomidine at a total dose of 0.5 micrograms/kg [8].

Group Q: Includes 63 women. Those patients will receive bilateral ultrasound-guided quadratus lumborum, lateral approach with a total volume of 60 ml of bupivacaine 0.3% and dexmedetomidine at a total dose of 0.5 mg/kg.

* Sample Size: Sample size was calculated using PASS II software. setting the type-1 error (α) at 0.05 , power (1-β) at 0.8 and confidence width level at 0.1 , Calculation according to the values of previous studies' Comparative efficacy of quadratus lumborum type II and erector spinae plane block in patients undergoing caesarean section under spinal anesthesia: a randomized controlled trial produced a sample size of at least 63 cases for each group.
* Ethical Considerations: The study will be conducted after approval by the Research Ethics Committee of the Faculty of Medicine, Ain Shams University, and conducted in accordance with the principles of the Declaration of Helsinki. A written informed consent before enrolment will be taken.
* Study Procedures:

All patients will be monitored at 2 hrs. postpartum and every 6 hrs. for 24 hours, and the following will be recorded: The need for adjuvant analgesics, the first time to ask for adjuvants, the beginning of the mother-baby bond, the ambulation of the patients, the pain score using a numerical analogue scale, the type of pain, if there is a change in SBP > 20 mmHg or HR > 20/min, an increase in RR > 10 above baseline or a 5% decrease in SaO2, and the time for discharge. The patient's satisfaction to the block will be measured using 4 points Likert assessment to the question, "Are you satisfied with the pain management done after the caesarean section?" totally disagree, disagree, Agree, totally agree. In case the patient feels pain after the block, it will be managed in a stepwise manner, and each step will be recorded by ketorolac (30 mg prn every 8 hr) and recorded. Paracetamol 1gm prn every 6hr and will be recorded. Morphine 4 mg incremental dose up to achieving the target level with a maximum dose 0.1 mg/kg/dose prn every 6 hrs. and will be recorded. The patient with failed block will be recorded and managed by the aforementioned steps, and the investigators will consider repeating the block. Failure of the block means that the patient is feeling severe agonizing pain that interferes with her physical and social activities, such as taking a normal breath, starting breastfeeding, starting movement, and so on.

• Statistical analysis All statistical procedures will be conducted using SPSS version 20 for Windows (SPSS Inc, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Parturient female
* Scheduled for elective cesarean section

Exclusion Criteria:

* Known allergy to any of the medications used
* Patients refused to participate in the study
* Patients with emergency section,
* Patients with Bleeding disease
* Patients with postpartum haemorrhage

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To test whether the type of the plane block have an implication on the patients' satisfaction. | first 24 hours after the surgery
  The patient's satisfaction with the block will be measured using a 4-point Likert assessment to the question, "Are you satisfied with the pain management done after the cesarean section?" totally disagree, disagree, agree, totally agree.

SECONDARY OUTCOMES:
to test the difference between the two approaches on the hospital discharge | 24-48 hours after the surgery
  report the time for discharge from the hospital after the surgery and if there is any delay or complications after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Wael S El Gharabawy, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Sutton CD, Carvalho B. Optimal Pain Management After Cesarean Delivery. Anesthesiol Clin. 2017 Mar;35(1):107-124. doi: 10.1016/j.anclin.2016.09.010. Epub 2016 Dec 12. PMID 28131114
- [Background] Wikner M. Unexpected motor weakness following quadratus lumborum block for gynaecological laparoscopy. Anaesthesia. 2017 Feb;72(2):230-232. doi: 10.1111/anae.13754. Epub 2016 Nov 28. PMID 27891579
- [Background] Ribeiro Junior IDV, Carvalho VH, Brito LGO. Erector spinae plane block for analgesia after cesarean delivery: a systematic review with meta-analysis. Braz J Anesthesiol. 2022 Jul-Aug;72(4):506-515. doi: 10.1016/j.bjane.2021.09.015. Epub 2021 Oct 18. PMID 34673125
- [Background] Priya TK, Singla D, Talawar P, Sharma RS, Goyal S, Purohit G. Comparative efficacy of quadratus lumborum type-II and erector spinae plane block in patients undergoing caesarean section under spinal anaesthesia: a randomised controlled trial. Int J Obstet Anesth. 2023 Feb;53:103614. doi: 10.1016/j.ijoa.2022.103614. Epub 2022 Dec 6. PMID 36535864
- [Background] Yu L, Shen X, Liu H. The effect and safety of dexmedetomidine as an adjuvant to local anesthetics in erector spinae plane block: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2023 Feb 27;23(1):61. doi: 10.1186/s12871-023-02019-x. PMID 36849910